CLINICAL TRIAL: NCT03911999
Title: To Investigate the Diagnostic Accuracy of Exosomal microRNA in Predicting the Aggressiveness of Prostate Cancer in Chinese Patients
Brief Title: Exosomal microRNA in Predicting the Aggressiveness of Prostate Cancer in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2018.063
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-prostate cancer subjects: No clinical evidence of prostate cancer
- Subjects with pathologically insignificant prostate cancer: Insignificant prostate cancers were organ confined with tumor volumes less than 0.5 cc and Gleason score < 7.
- Subjects with pathologically significant prostate cancer: Significant cancers are those with either Gleason score > 7, evidences of extra-prostatic extension with positive margins, or seminal vesicles / lymph nodes involvement.

SUMMARY:
The prostate gland is a clinically important male accessory sex gland and vital for its production of semen. Prostate cancer (PCa) is now ranked 3th in annual incidence of male cancer and ranked 5th for cancer-related death in men in Hong Kong which accounts for about 10.9 deaths per 100,000 persons. Its incidence is rising rapidly, almost tripled in the past 10 years. Fortunately, with the improvement in awareness of the disease and also increasing use of serum prostate specific antigen for early case identification, many patients are diagnosed at an earlier stage. However, unlike other malignancy, PCa is characterized by its slow progression nature. Therefore, some patients with low grade low volume disease might never suffered from PCa related complications or mortality. As a result, recent year, there is an increase use a more conservative approach, active surveillance (AS), for management of early prostate cancer. The principle of AS is selecting patients with low risk of disease and offered them regular monitoring, instead of radical local therapy, unless patient's cancer was noticed to progressing. By using this approach, patients might avoid possible complications related to treatment. Currently, people could use some clinical parameters, imaging and repeated prostate biopsy to assess and monitor the aggressiveness/ progression of PCa. However, these parameters suffered from defects, such as low correlation to the final PCa pathology or not readily repeatable for patients. Therefore, there is a need to identify more easy, safe and repeatable monitoring of the aggressiveness of prostate cancer.

Exosome is genetic materials secreted by cells and could be measured in various body fluid. There are some studies suggested it is a potential marker for PCa diagnosis and monitoring. The aim of this study is to investigate the relationship of urinary exosome and the aggressiveness of prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the third most common male cancer in Hong Kong. While the use of serum PSA has greatly improved the proportion of patients diagnosed at localized /early stage, there are also problems of overdiagnosis and overtreatment. Unfortunately, there was still no ideal markers that could help to predict the aggressiveness of PCa, especially in Chinese population. Exosome is an important media for cell-cell interaction. The content of exomsomes, including microRNAs, are believed to have important roles in PCa development and progression, and might also serve as potential markers in PCa management. Therefore, investigators would like to explore the role of exosomal microRNA in the prediction of tumour aggressiveness in local Chinese PCa patients. This is a prospective study divided into two parts. Subjects will be recruited consecutively from two hospitals.

In Part I of the study (Candidate exosomal microRNA discovery and selection), a total of 60 patients from three groups (non-cancer, pathologically insignificant cancer and significant cancer patients) will be recruited. First portion of urine will be collected from them. For Group 2&3 patients, they are patients with clinically localized prostate cancer and planned for radical prostatectomy, urine will be collected before surgery for these two groups. Exosomal RNA will be extracted from urine and microRNAs expression profiles will be determined by next-generation sequencing. Candidate exosomal microRNAs that could differentiate pathological insignificant and significant PCa will be identified for Part II study.

In Part II study (Candidate exosomal microRNAs validation), 180 patients with localized prostate cancer, planned for radical prostatectomy will be recruited. Urine will be again collected before surgery and the level of candidate exosomal microRNAs for each patient will be assessed. The diagnostic accuracy of these candidate exosomal microRNAs on predicting pathological insignificant cancer and also correlation with the final pathology will be assessed.

The primary tasks for Part I study is the identification of potential exosomal microRNAs that could differentiate pathologically insignificant and significant PCa.

The primary task for Part II study is the validation of the ability of those candidate exosomal microRNAs in differentiating pathological insignificant and significant PCa.

ELIGIBILITY:
Inclusion Criteria:

1. For non prostate cancer group

   * Male subject with age 45 or above
   * No clinical evidence of PCa, serum PSA <4 ng/dl and normal digital rectal examination.
2. For prostate cancer group

   * Male subject with age 45 or above
   * Clinically diagnosed to have localized PCa and planned for radical prostatectomy
   * No prior systemic therapy for PCa used, including hormonal or chemotherapy.

Exclusion Criteria:

* History of medications usage that can affect serum PSA levels within 6 months of study enrolment.
* History of active urinary tract infection within 1 month of study enrolment.
* History of invasive prostate / bladder treatments within 6 months of study enrolment.
* History of concurrent renal/bladder cancer within 6 months of study enrolment.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For non prostate cancer group, there is no specific time limit for urine collection. For prostate cancer group, urine will be collected prior to prostatectomy.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
To compare the differences in microRNA expression between non-prostate cancer subjects, pathologically insignificant and significant prostate cancer patients. | Baseline, one-time point
  Urine will be collected prior to surgery. The urine sample will then be handled immediately for exosomal RNA extraction (refer to specific methodology). The extracted exosomal RNA would then be stored for next generation sequencing (NGS). Results of the 3 groups will then be compared, with reference to literatures findings. Candidate microRNAs that can differentiate between pathologically significant and insignificant cancer will be selected for Part II study.
To assess the accuracy of selected microRNAs for the differentiation of patients with pathologically insignificant and significant prostate cancer after radical prostatectomy | Baseline, one-time point
  Urine will be collected prior to surgery. The urine sample will then be handled immediately for exosomal RNA extraction (refer to specific methodology). The extracted exosomal RNA would then be stored for next generation sequencing (NGS). Results of the 3 groups will then be compared, with reference to literatures findings. Candidate microRNAs that can differentiate betten pathologically significant and insignificant cancer will be selected for Part II study.The preoperative patients and disease parameters, including age, clinical staging, serum PSA level, prostatic biopsy results, MRI findings, together with the prostatectomy pathology will be collected for subsequent data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Strope SA, Andriole GL. Prostate cancer screening: current status and future perspectives. Nat Rev Urol. 2010 Sep;7(9):487-93. doi: 10.1038/nrurol.2010.120. PMID 20818326
- [Background] Epstein JI, Walsh PC, Carmichael M, Brendler CB. Pathologic and clinical findings to predict tumor extent of nonpalpable (stage T1c) prostate cancer. JAMA. 1994 Feb 2;271(5):368-74. PMID 7506797
- [Background] Ploussard G, Epstein JI, Montironi R, Carroll PR, Wirth M, Grimm MO, Bjartell AS, Montorsi F, Freedland SJ, Erbersdobler A, van der Kwast TH. The contemporary concept of significant versus insignificant prostate cancer. Eur Urol. 2011 Aug;60(2):291-303. doi: 10.1016/j.eururo.2011.05.006. Epub 2011 May 17. PMID 21601982
- [Background] McKiernan J, Donovan MJ, O'Neill V, Bentink S, Noerholm M, Belzer S, Skog J, Kattan MW, Partin A, Andriole G, Brown G, Wei JT, Thompson IM Jr, Carroll P. A Novel Urine Exosome Gene Expression Assay to Predict High-grade Prostate Cancer at Initial Biopsy. JAMA Oncol. 2016 Jul 1;2(7):882-9. doi: 10.1001/jamaoncol.2016.0097. PMID 27032035
- [Background] Dinh KT, Mahal BA, Ziehr DR, Muralidhar V, Chen YW, Viswanathan VB, Nezolosky MD, Beard CJ, Choueiri TK, Martin NE, Orio PF, Sweeney CJ, Trinh QD, Nguyen PL. Incidence and Predictors of Upgrading and Up Staging among 10,000 Contemporary Patients with Low Risk Prostate Cancer. J Urol. 2015 Aug;194(2):343-9. doi: 10.1016/j.juro.2015.02.015. Epub 2015 Feb 11. PMID 25681290
- [Background] Chiu PK, Lai FM, Teoh JY, Lee WM, Yee CH, Chan ES, Hou SM, Ng CF. Prostate Health Index and %p2PSA Predict Aggressive Prostate Cancer Pathology in Chinese Patients Undergoing Radical Prostatectomy. Ann Surg Oncol. 2016 Aug;23(8):2707-14. doi: 10.1245/s10434-016-5183-6. Epub 2016 Mar 10. PMID 26965697
- [Background] Schiffer E. Biomarkers for prostate cancer. World J Urol. 2007 Dec;25(6):557-62. doi: 10.1007/s00345-007-0203-6. Epub 2007 Aug 10. PMID 17690889
- [Background] Ng CF, Yeung R, Chiu PK, Lam NY, Chow J, Chan B. The role of urine prostate cancer antigen 3 mRNA levels in the diagnosis of prostate cancer among Hong Kong Chinese patients. Hong Kong Med J. 2012 Dec;18(6):459-65. PMID 23223645
- [Background] Laxman B, Tomlins SA, Mehra R, Morris DS, Wang L, Helgeson BE, Shah RB, Rubin MA, Wei JT, Chinnaiyan AM. Noninvasive detection of TMPRSS2:ERG fusion transcripts in the urine of men with prostate cancer. Neoplasia. 2006 Oct;8(10):885-8. doi: 10.1593/neo.06625. PMID 17059688
- [Background] Ren S, Peng Z, Mao JH, Yu Y, Yin C, Gao X, Cui Z, Zhang J, Yi K, Xu W, Chen C, Wang F, Guo X, Lu J, Yang J, Wei M, Tian Z, Guan Y, Tang L, Xu C, Wang L, Gao X, Tian W, Wang J, Yang H, Wang J, Sun Y. RNA-seq analysis of prostate cancer in the Chinese population identifies recurrent gene fusions, cancer-associated long noncoding RNAs and aberrant alternative splicings. Cell Res. 2012 May;22(5):806-21. doi: 10.1038/cr.2012.30. Epub 2012 Feb 21. PMID 22349460
- [Background] Gudmundsson J, Sulem P, Gudbjartsson DF, Masson G, Agnarsson BA, Benediktsdottir KR, Sigurdsson A, Magnusson OT, Gudjonsson SA, Magnusdottir DN, Johannsdottir H, Helgadottir HT, Stacey SN, Jonasdottir A, Olafsdottir SB, Thorleifsson G, Jonasson JG, Tryggvadottir L, Navarrete S, Fuertes F, Helfand BT, Hu Q, Csiki IE, Mates IN, Jinga V, Aben KK, van Oort IM, Vermeulen SH, Donovan JL, Hamdy FC, Ng CF, Chiu PK, Lau KM, Ng MC, Gulcher JR, Kong A, Catalona WJ, Mayordomo JI, Einarsson GV, Barkardottir RB, Jonsson E, Mates D, Neal DE, Kiemeney LA, Thorsteinsdottir U, Rafnar T, Stefansson K. A study based on whole-genome sequencing yields a rare variant at 8q24 associated with prostate cancer. Nat Genet. 2012 Dec;44(12):1326-9. doi: 10.1038/ng.2437. Epub 2012 Oct 28. PMID 23104005
- [Background] Wang G, Chan ES, Kwan BC, Li PK, Yip SK, Szeto CC, Ng CF. Expression of microRNAs in the urine of patients with bladder cancer. Clin Genitourin Cancer. 2012 Jun;10(2):106-13. doi: 10.1016/j.clgc.2012.01.001. Epub 2012 Mar 3. PMID 22386240
- [Background] Kumar B, Lupold SE. MicroRNA expression and function in prostate cancer: a review of current knowledge and opportunities for discovery. Asian J Androl. 2016 Jul-Aug;18(4):559-67. doi: 10.4103/1008-682X.177839. PMID 27056344
- [Background] Endzelins E, Melne V, Kalnina Z, Lietuvietis V, Riekstina U, Llorente A, Line A. Diagnostic, prognostic and predictive value of cell-free miRNAs in prostate cancer: a systematic review. Mol Cancer. 2016 May 18;15(1):41. doi: 10.1186/s12943-016-0523-5. PMID 27189160
- [Background] Yu S, Wang X, Ng CF, Chen S, Chan FL. ERRgamma suppresses cell proliferation and tumor growth of androgen-sensitive and androgen-insensitive prostate cancer cells and its implication as a therapeutic target for prostate cancer. Cancer Res. 2007 May 15;67(10):4904-14. doi: 10.1158/0008-5472.CAN-06-3855. PMID 17510420
- [Background] Tsoi TH, Chan CF, Chan WL, Chiu KF, Wong WT, Ng CF, Wong KL. Urinary Polyamines: A Pilot Study on Their Roles as Prostate Cancer Detection Biomarkers. PLoS One. 2016 Sep 6;11(9):e0162217. doi: 10.1371/journal.pone.0162217. eCollection 2016. PMID 27598335
- [Background] Zhang DZ, Lau KM, Chan ES, Wang G, Szeto CC, Wong K, Choy RK, Ng CF. Cell-free urinary microRNA-99a and microRNA-125b are diagnostic markers for the non-invasive screening of bladder cancer. PLoS One. 2014 Jul 11;9(7):e100793. doi: 10.1371/journal.pone.0100793. eCollection 2014. PMID 25014919
- [Background] Leung YK, Chan QK, Ng CF, Ma FM, Tse HM, To KF, Maranchie J, Ho SM, Lau KM. Hsa-miRNA-765 as a key mediator for inhibiting growth, migration and invasion in fulvestrant-treated prostate cancer. PLoS One. 2014 May 16;9(5):e98037. doi: 10.1371/journal.pone.0098037. eCollection 2014. PMID 24837491